CLINICAL TRIAL: NCT00302120
Title: MR Mammography: Randomized Controlled Trial to Study Efficiency of MR Mammography in Reducing the Number of Invasive Interventions in Nonpalpable Suspicious Breast Lesions. The MONET - Study
Brief Title: The MONET - Study: MR Mammography of Nonpalpable Breast Tumors
Acronym: MONET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Porf. dr. W. Mali / Prof. dr. P. Peeters, University Medical Center Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UMC Utrecht
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Breast Neoplasms
Keywords: Magnetic Resonance Imaging; Breast Neoplasms; Diagnostic Trial
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: Contrast-enhanced MR mammography

SUMMARY:
The purpose of this study is to determine whether performing MRI of the breast will improve breast cancer management by reducing the number of biopsies and in case of malignancy allowing one-stage surgical excision of the tumor.

DETAILED DESCRIPTION:
Each year 7000 women present with nonpalpable suspicious breast lesions on mammography in the Netherlands. In the usual care situation, these lesions are detected by mammography and ultrasonography and pathologically characterized by analysis of large core needle biopsy material. In case of malignancy, these lesions are surgically removed. First, a wire is placed in the breast with the tip of the wire within 1 cm of the tumor and then the surgeon follows the wire and removes the lesion. Unfortunately about 25% of women require more that one surgical procedure to remove all tumorous tissue. This is caused by incorrect presurgical diagnosis of the extent and invasiveness of the disease (multifocality, multicentricity, lymph node involvement). We hypothesize that MR mammography will improve presurgical diagnosis and differentiation of lesions and thereby decrease the number of invasive surgical procedures (primary outcome) and number of invasive biopsies (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* patients with a nonpalpable, mammographically suspicious breast lesion (BI-RADS 3, 4 or 5)
* referred for large core needle biopsy
* 18 to 75 years

Exclusion Criteria:

* previous breast surgery or radiation therapy of the breast less than 9 months before MR mammography
* pregnant or lactating
* claustrophobia or adiposity ( > 130 kg)
* general contraindications for MRI
* unable to maintain prone position for one hour
* medically unstable patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The absolute number of surgical procedures in women with nonpalpable malignancies will be compared between MRI group and control group. | 2010

SECONDARY OUTCOMES:
The number of large core needle biopsies that can be prevented because of a definite diagnosis as provided by MRI will be calculated. | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Willem P Mali, MD PhD, Study Director — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Meander Medisch Centrum, Amersfoort
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Unicersity Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Peters NH, Borel Rinkes IH, Mali WP, van den Bosch MA, Storm RK, Plaisier PW, de Boer E, van Overbeeke AJ, Peeters PH. Breast MRI in nonpalpable breast lesions: a randomized trial with diagnostic and therapeutic outcome - MONET - study. Trials. 2007 Nov 28;8:40. doi: 10.1186/1745-6215-8-40. PMID 18045470